CLINICAL TRIAL: NCT05647616
Title: Strengthening of the Peroneus Longus Muscle in Patients With Dorsiflexed First Ray
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Pedro V. Munuera-Martínez, Profesor Titular de Universidad, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Peroneus Longus and First Ray
Record Dates: First submitted 2022-12-02; First posted 2022-12-12 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: First Ray Dorsiflexion

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strengthening exercises (Experimental): The participants in this group will be given instructions to follow a resistance exercises to strengthen the peroneus longs muscle.
  Interventions: Other: Strengthening exercises
- Control (No Intervention): Participants in this group will be given no treatment.

INTERVENTIONS:
Other: Strengthening exercises — Participants in group A will be required to complete 12 sessions in 4 to 6 weeks. Resistance-Bands will be used to do ankle plantar flexion and eversion (3 sets of 10 repetitions). Participants will have to be seated on the floor with the knee extended and instructed to perform the movement at the ankle joint without allowing extraneous movement at hip and knee. The resistance band will be doubled and securely attached to the base of a table. The training resistance will be determined by calculating 70% of the resting length of the resistance band and adding this distance to the resting length of the resistance band. Using this calculated distance, the examiner will place a mark to which the resistance band will be stretched during exercise performance on the floor. Each week a study investigator will track each participant's completion. Participants will be instructed to move through their entire range of motion for the direction of each exercise.
  Arms: Strengthening exercises

SUMMARY:
BACKGROUND: The first metatarsal and medial cuneiform form an important functional unit in the foot called "first ray". The first ray normal function requires that it load part of the body weight in the last period of the stance phase of gait. A dorsiflexed first ray may exist due to abnormal function of the peroneus longus muscle.

OBJECTIVE: To evaluate the improvement in first ray function in tha push-off phase of gait after a 4-week strengthening programme for the peroneus longus.

SUBJECTS: Patients with flexible dorsiflexed first ray. INTERVENTIONS: Patients will be randomly assigned to either group A, which will receive instructions for a strengthening programme of the peroneus longus muscle, or group B, which will receive no treatment.

MAIN MEASURES: The primary outcomes will be mean and maximum plantar pressure under the first metatarsal head.

ELIGIBILITY:
Inclusion Criteria:

* Flexible dorsiflexed first ray.

Exclusion Criteria:

* Traumatisms on the feet in the last 12 months.
* Previous foot surgery.
* Hallux abducto-valgus.
* Being in treatment with foot orthoses.
* Systemic musculoskeletal disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum plantar pressure under the first metatarsal head | Four weeks
  The maximum plantar pressure detected by a pressure plate with capacitive sensors under the first metatarsal head load area.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro V Munuera-Martínez, Ph.D, Study Director — University of Seville
Locations (1):
- Department of Podiatry, Seville, Spain

IPD SHARING:
Plan to Share IPD: No